CLINICAL TRIAL: NCT03497689
Title: EXPEDITE: A 16-Week, Multicenter, Open-label Study of Remodulin Induction Followed by Orenitram Optimization in Subjects With Pulmonary Arterial Hypertension
Brief Title: EXPEDITE: A Study of Remodulin Induction Followed by Orenitram Optimization to Treat Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-402
Record Dates: First submitted 2018-03-20; First posted 2018-04-13 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary hypertension; Treprostinil; Pulmonary arterial hypertension; Remodulin; Orenitram
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous/Subcutaneous Treprostinil; Oral Treprostinil (Experimental): Subjects began Remodulin at 2 ng/kg/min subcutaneously (SC) or intravenously (IV) and were optimized to their maximum tolerated dose (MTD) of Remodulin. Subjects were then transitioned to Orenitram XR tablets (oral) based upon their Remodulin dose. Subjects were optimized on Orenitram therapy to a MTD. There were no maximum Remodulin or Orenitram doses specified during the study.
  Interventions: Drug: Intravenous/Subcutaneous Treprostinil; Oral Treprostinil

INTERVENTIONS:
Drug: Intravenous/Subcutaneous Treprostinil; Oral Treprostinil — Short-term course of IV or SC treprostinil continuous infusion followed by transition to oral treprostinil extended-release (XR) tablets taken 3 times daily (TID)
  Other Names: Remodulin; Orenitram

SUMMARY:
This was a multicenter, open-label study to evaluate the dose of Orenitram® (treprostinil) Extended Release Tablets achieved at 16 weeks after a short-term course of Remodulin® (treprostinil) Injection in subjects with pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
Subjects were initiated on subcutaneous (SC) or intravenous (IV) treprostinil and titrated to a dose that improved the symptoms of PAH while minimizing excessive pharmacologic effects. After achieving a minimum SC/IV treprostinil dose of 20 ng/kg/min, subjects began a transition to oral treprostinil at the Transition Visit, which occurred at the Week 2, 4, or 8 study visit. After the Transition Visit, oral treprostinil titration continued through Week 16 to reach the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntary gave written informed consent to participate in study.
2. Males and female subjects aged 18 to 75 years at Screening (date the subject provided written informed consent to participate in study).
3. Subjects with a diagnosis of World Health Organization (WHO) Group 1 pulmonary hypertension (PH): symptomatic idiopathic or heritable PAH; or PAH associated with connective tissue disease, human immunodeficiency virus (HIV) infection, repaired congenital systemic-to-pulmonary shunt (at least 1 year since repair with respect to the date of providing informed consent), or appetite suppressant/toxin use.
4. Subjects with WHO functional class (FC) II or III symptoms at Baseline.
5. Subjects with 6MWD >250 m at Baseline.
6. Subjects who were either not receiving PAH-targeted therapy or were currently being treated with 1 or 2 oral FDA-approved PAH therapies consisting of an endothelin receptor antagonist (ERA) and/or either a phosphodiesterase type-5 inhibitor (PDE5-I) or a soluble guanylate cyclase (sGC) stimulator for ≥45 days, and on a stable dose for ≥30 days prior to the Baseline Visit.
7. Subjects on stable doses of other medical therapies for at least 10 days prior to the Baseline Visit, with no dose adjustments, additions, or discontinuations, with the exception of discontinuation or dose changes of anticoagulants and/or diuretics. Subjects could not have recent changes to non-pharmacologic interventions, such as exercise, diet plans, pulmonary rehabilitation, or sleep apnea treatment, for at least 10 days prior to Baseline Visit.
8. Subjects with historical right heart catheterization (RHC) results consistent with WHO Group 1 PH, as demonstrated by pulmonary artery pressure mean of ≥25 mmHg, a pulmonary artery wedge pressure (PAWP) or left ventricular (LV) end-diastolic pressure ≤15 mmHg (if a PAWP measurement was not available) and a pulmonary vascular resistance (PVR) >3 Wood units, in the absence of unrepaired congenital heart disease (other than patent foramen ovale).
9. Subject underwent an RHC within 180 days of Baseline and had a cardiac index ≥2.0 L/min/m² with no changes in their PAH medication regimen (ie, both dosing and drug) since the RHC.
10. Subjects with most recent historical echocardiogram (ECHO) demonstrating clinically normal left systolic and diastolic ventricular function and absence of any clinically significant left-sided heart disease. Subjects with clinically insignificant LV diastolic dysfunction due to the effects of right ventricular (RV) overload (RV hypertrophy and/or RV dilation) were eligible.
11. Subjects who agreed to follow the specified precautions to avoid pregnancy as follows:

    1. For female subjects of childbearing potential, a negative urine pregnancy test was required at Screening and Baseline prior to initiating study drug. Female subjects of childbearing potential must have followed 1 of the following approaches: i. practice actual abstinence from intercourse, ii. had a partner with a vasectomy, iii. had an intrauterine device, or iv. must have used 2 different forms of highly effective contraception for the duration of the study, and for at least 48 hours after discontinuing study drug. Medically acceptable forms of effective contraception included approved hormonal contraceptives (such as birth control pills) or barrier methods (such as a condom or diaphragm).
    2. Male subjects with a partner of childbearing potential must have used a condom during intercourse for the duration of the study, and for 48 hours after discontinuing study drug.
12. HIV-positive subjects must have had a CD4 lymphocyte count of at least 200 cells/mm^3 within 30 days of Screening and been receiving current standard-of-care anti-retroviral or other effective medication for the treatment of HIV, with no changes for at least 8 weeks prior to enrollment.
13. Subjects who, in the opinion of the Investigator, were capable of communicating effectively with study personnel and were considered reliable, willing, and likely to be cooperative with protocol requirements and attend all required study visits.
14. Subjects who had the capability to answer surveys and questionnaires written in English.

Exclusion Criteria:

1. Female subjects who were pregnant, lactating, or planning to become pregnant during the study.
2. Subjects with a current diagnosis of uncontrolled sleep apnea, as defined by their physician.
3. Subjects with renal insufficiency, as defined by requiring dialysis or an estimated creatinine clearance of <30 mL/min, as calculated by the Cockcroft-Gault equation.
4. Subjects with liver dysfunction defined as elevated liver function tests (alanine aminotransferase or aspartate aminotransferase) ≥3 times the upper limit of normal at Screening, or subjects with Child-Pugh Class B or C hepatic disease.
5. Subjects with anemia, as defined by Screening hemoglobin <9 g/dL.
6. Subjects with an active infection or condition that interfered with interpretation of study assessments.
7. Subjects with a history of ischemic heart disease (defined as subjects who required anti-anginal therapy within 6 months of Screening or who had experienced a documented myocardial infarction within 6 months of Screening) or a history of left-sided myocardial dysfunction, as evidenced by a PAWP >15 mmHg or LV ejection fraction <50%.
8. Subjects with uncontrolled systemic hypertension, as evidenced by systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg at Baseline.
9. Subjects with severe hypotension, as evidenced by systolic blood pressure <90 mmHg or diastolic blood pressure <50 mmHg at Baseline.
10. If a lung assessment was completed as per standard of care, any subject with 1 or more of the following signs of documented relevant lung disease within 180 days of Baseline: total lung capacity <60% of predicted or forced expiratory volume in 1 second <55% of predicted normal.
11. Subjects with chronic musculoskeletal disorder or any other disease that limited ambulation, or who were connected to a machine that was not portable.
12. Subjects with a history of alcohol abuse or illicit drug abuse within 12 months of Baseline which, in the Investigator's opinion, made the subject inappropriate for enrollment in a clinical study.
13. Subjects with any other concomitant disease with life expectancy of <12 months from Baseline.
14. Subjects with an unstable psychiatric condition or those not capable of understanding the objectives, nature, or consequences of the study, or who have any condition which, in the Investigator's opinion, constituted an unacceptable risk to the subject's safety.
15. Subjects who were currently receiving an investigational drug, had an investigational device in place, or who had participated in an investigational drug or device study within 180 days prior to Baseline. Participation in an observational study within 180 days prior to Baseline did not disqualify a subject from enrolling.
16. Subjects who had received a prostacyclin-class therapy within 28 days of Baseline.
17. Subjects who had a Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) 2.0 Risk Score of ≥10.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Miller, MD, Principal Investigator — Piedmont Healthcare Pulmonary and Critical Care Research
Locations (11):
- United States (11):
  - University of California San Francisco - Fresno, Fresno, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Florida Hospital, Orlando, Florida
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Cincinnati Health, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - UPMC Presbytarian Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller CE, Franco V, Smith JS, Balasubramanian V, Kingrey J, Zolty R, Melendres-Groves L, Huston J, Elwing JM, Ravichandran A, Cella D, Shen E, Seaman S, Thrasher CM, Broderick M, Oudiz RJ. Parenteral treprostinil induction for rapid attainment of therapeutic doses of oral treprostinil. Respir Med. 2023 Nov;218:107374. doi: 10.1016/j.rmed.2023.107374. Epub 2023 Aug 1. PMID 37532157

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 36 subjects enrolled but only 35 subjects started treatment with Remodulin (Safety Population). One subject was enrolled but did not receive study drug due to a violation of entry criteria (CD4 lymphocyte count for HIV-positive subjects).
Groups:
- Intravenous/Subcutaneous Treprostinil; Oral Treprostinil: IV or SC treprostinil induction followed by transition to oral treprostinil
  Intravenous/Subcutaneous Treprostinil; Oral Treprostinil: Short-term course of IV or SC treprostinil continuous infusion followed by transition to oral treprostinil XR tablets taken TID
Period: Overall Study
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Started | 35
Completed | 28
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Intravenous/Subcutaneous Treprostinil; Oral Treprostinil: IV or SC treprostinil induction followed by transition to oral treprostinil
  Intravenous/Subcutaneous Treprostinil; Oral Treprostinil: Short term course of IV/SC treprostinil continuous infusion followed by transition to oral treprostinil extended-release (XR) tablets taken three times daily (TID)
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 56.0 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 29
  More than one race | 0
  Unknown or Not Reported | 1
PAH Etiology [Count of Participants; unit: Participants]
  Idiopathic PAH | 15
  Associated with connective tissue disease | 9
  Associated with appetite suppressant or toxin use | 7
  Associated with HIV infection | 1
  Heritable PAH | 1
  Other | 2
  Associated with repaired congenital systemic-to-pulmonary shunts | 0
Days Since Initial PAH Diagnosis [Median (Full Range); unit: days] | 245.0 [7 to 1959]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Oral Treprostinil Dose
Description: The number of subjects that achieved an oral treprostinil dose of ≥4 mg TID (or a total daily dose [TDD] of 12 mg) at Week 16 (or a dose of ≥0.057 mg/kg TID [TDD of 0.171 mg/kg] for subjects <70 kg).
Time Frame: Assessed at Week 16
Population: Per-protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 29
Participants | 23

2. Secondary Outcome: Change in 6-minute Walk Distance (6MWD)
Description: The 6-Minute Walk Test (6MWT) is used to measure exercise ability in patients with chronic respiratory diseases. The distance walked on a predetermined course over 6 minutes was recorded.
Time Frame: From Baseline to Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: meters
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 27
meters | 25.00 [-210.0 to 112.0]

3. Secondary Outcome: Change in Borg Dyspnea Score
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (no shortness of breath) to 10 (worst shortness of breath you have ever had).
Time Frame: From Baseline to Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 27
score on a scale | -1.00 [-5.0 to 4.0]

4. Secondary Outcome: Number of Subjects With Changes in WHO FC
Description: WHO FC ranges from I (subjects with PH but without resulting limitation of physical activity) to IV (subjects with PH with inability to carry out any physical activities without symptoms). A lower WHO FC was considered "improved"; a higher WHO FC was considered "worsened."
Time Frame: From Baseline to Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 28
Participants
  Improved | 19
  Worsened | 1
  No Change | 8

5. Secondary Outcome: Change in Serum N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Levels
Description: NT-proBNP is a hormone produced by the heart. NT-proBNP concentration is associated with changes in right heart morphology and function. The main purpose of NT-proBNP testing is to see if the blood levels of this protein are within the expected range for a healthy person. Normal levels of NT-proBNP are less than 125 pg/mL for people under 75 years old and less than 450 pg/mL for people over age 75. NT-proBNP levels over 900 pg/mL may be a sign of heart failure. The higher the level, the more serious the condition.
Time Frame: From Baseline to Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: ng/L
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 28
ng/L | -134.0 [-3896 to 556]

6. Secondary Outcome: Change in Echocardiogram Parameters (Change in Cardiac Output)
Description: ECHOs provide information regarding cardiac structure and function. Cardiac output was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: L/min
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
L/min | 0.55 [-1.7 to 3.1]

7. Secondary Outcome: Change in Echocardiogram Parameters (Heart Rate)
Description: ECHOs provide information regarding cardiac structure and function. Heart rate was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: beats/min
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
beats/min | 1.50 [-17.0 to 23.0]

8. Secondary Outcome: Change in Echocardiogram Parameters (Left Ventricular Outflow Track Dimension)
Description: ECHOs provide information regarding cardiac structure and function. Left ventricular outflow track (LVOT) dimension was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: mm
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 23
mm | 0.42 [-1.1 to 2.6]

9. Secondary Outcome: Change in Echocardiogram Parameters (LVOT Velocity Time Integral)
Description: ECHOs provide information regarding cardiac structure and function. LVOT velocity time integral was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: cm
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
cm | 0.93 [-6.8 to 7.7]

10. Secondary Outcome: Change in Echocardiogram Parameters (LV Diameter)
Description: ECHOs provide information regarding cardiac structure and function. LV diameter was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: mm
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 21
mm | 3.52 [-4.4 to 14.1]

11. Secondary Outcome: Change in Echocardiogram Parameters (LV Eccentricity Index [Diastole])
Description: ECHOs provide information regarding cardiac structure and function. LV Eccentricity Index (Diastole) was summarized at each time point listed. Diastole LV Eccentricity Index is measured during ECHOs to assess how much the shape of the LV deviates from normal while the heart is relaxing (full of blood prior to contraction). A lower Diastole LV Eccentricity Index indicates that the LV is closer to a normal shape during diastole. A higher Diastole LV Eccentricity Index indicates that the LV is more elongated/stretched during diastole, indicating potential heart problems. There is no theoretical minimum or maximum value for the index range.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: Eccentricity Index
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
Eccentricity Index | 0.04 [-0.3 to 0.3]

12. Secondary Outcome: Change in Echocardiogram Parameters (LV Eccentricity Index [Systole])
Description: ECHOs provide information regarding cardiac structure and function. LV Eccentricity Index (Systole) was summarized at each time point listed. Systole LV Eccentricity Index is measured during ECHOs to assess how much the shape of the LV deviates from normal while the heart is contracting (pumping blood to the body). A lower Systole LV Eccentricity Index indicates that the LV is closer to a normal shape during systole. A higher Systole LV Eccentricity Index indicates that the LV is more elongated/stretched during systole, indicating potential heart problems. There is no theoretical minimum or maximum value for the index range.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: Eccentricity Index
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
Eccentricity Index | 0.09 [-1.0 to 0.7]

13. Secondary Outcome: Change in Echocardiogram Parameters (Pulmonary Valve Acceleration Time)
Description: ECHOs provide information regarding cardiac structure and function. Pulmonary valve acceleration time was summarized at each time point listed.=.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: msec
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 20
msec | 4.43 [-22.0 to 41.2]

14. Secondary Outcome: Change in Echocardiogram Parameters (RV/LV Ratio)
Description: ECHOs provide information regarding cardiac structure and function. RV/LV (diastole) ratio was summarized at each time point listed. RV/LV Ratio is the ratio of right ventricular to left ventricular diameter. A normal RV/LV Ratio is 0.6 to 1.0. When the ratio exceeds 1.0 it is indicative of high pulmonary artery pressure or right ventricular hypertrophy.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: Ratio
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 20
Ratio | -0.6 [-0.6 to 0.3]

15. Secondary Outcome: Change in Echocardiogram Parameters (Right Atrial Area)
Description: ECHOs provide information regarding cardiac structure and function. Right atrial area was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: cm^2
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 23
cm^2 | -2.88 [-15.8 to 5.3]

16. Secondary Outcome: Change in Echocardiogram Parameters (RV Diameter)
Description: ECHOs provide information regarding cardiac structure and function. RV diameter was summarized at each time point.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: mm
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 20
mm | -2.61 [-16.6 to 18.8]

17. Secondary Outcome: Change in Echocardiogram Parameters (RV Free Wall Strain)
Description: ECHOs provide information regarding cardiac structure and function. RV free wall strain was summarized at each time point listed .
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: percent
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 18
percent | 1.28 [-8.2 to 15.4]

18. Secondary Outcome: Change in Echocardiogram Parameters (RV Myocardial Performance Index)
Description: ECHOs provide information regarding cardiac structure and function. RV myocardial performance index (MPI) was summarized at each time point listed. RV MPI is a measurement used to assess RV systolic function in patients with PH. MPI correlates with pulmonary arterial pressure. Normal MPI is approximately 0.35. Higher MPI values indicate higher pulmonary arterial pressure.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: MPI
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
MPI | -0.08 [-0.6 to 0.5]

19. Secondary Outcome: Change in Echocardiogram Parameters (Tricuspid Annular Plane Systolic Excursion)
Description: ECHOs provide information regarding cardiac structure and function. Tricuspid annular plane systolic excursion was summarized at each time point listed.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: mm
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 22
mm | 1.20 [-5.0 to 7.8]

20. Secondary Outcome: Change in PAH Symptom Score
Description: PAH symptoms included fatigue, dyspnea, lower extremity edema, dizziness, syncope, chest pain, and orthopnea. Symptoms were scored (Grades 0 [none], 1 [mild], 2 [moderate], to 3 [severe]) except for syncope (0 [No], 1 [Infrequent; 1 episode], 2 [Somewhat frequent; 2 to 3 episodes], and 3 [Often; >4 episodes). A lower score was considered "improved"; a higher score was considered "worsened."
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. The Count of Participants analyzed in each row differs from the Overall Number of Participants since only subjects with Baseline and Week 16 values were measured and analyzed (ie, contributed data reported in the table).
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 28
Participants
  Fatigue: Improved | 11
  Fatigue: Worsened | 3
  Fatigue: No Change | 14
  Dyspnea: Improved | 17
  Dyspnea: Worsened | 1
  Dyspnea: No Change | 10
  Lower Extremity Edema: Improved | 8
  Lower Extremity Edema: Worsened | 4
  Lower Extremity Edema: No Change | 16
  Dizziness: Improved | 7
  Dizziness: Worsened | 4
  Dizziness: No Change | 17
  Syncope: Improved | 1
  Syncope: Worsened | 1
  Syncope: No Change | 26
  Chest Pain: Improved | 3
  Chest Pain: Worsened | 2
  Chest Pain: No Change | 23
  Orthopnea: Improved | 8
  Orthopnea: Worsened | 2
  Orthopnea: No Change | 18

21. Secondary Outcome: Change in Patient-reported Outcomes (Health-related Quality of Life)
Description: The Health-related Quality of Life in Pulmonary Hypertension Questionnaire (emPHasis-10) is a 10-question questionnaire used during clinical assessments that measures quality of life by the patients participating in the study. The patients graded their response to each of the 10 health-related questions on a scale of 0 to 5 based on how they were feeling that day. The most favorable score for each question is 0, and the least favorable score for each question is 5. A total score was then summed for each subject based on their responses to the 10 questions. The lower the total score was (best possible total score was 0), the less living with PH was negatively affecting the quality of the patient's life. The higher the total score (worst possible score was 50), the more living with PH was negatively affecting the quality of the patient's life.
Time Frame: At Baseline and Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 27
score on a scale | -3.0 [-33 to 16]

22. Secondary Outcome: Change in Treatment Satisfaction
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) is a 14-question questionnaire that measures the level of satisfaction or dissatisfaction patients have with their study medication in 4 areas: effectiveness (3 questions), side effects (5 questions), convenience (3 questions), and global satisfaction (3 questions). With the exception of the first side effects question (a yes or no question), all items have 5 or 7 responses which are scored from 1 (least satisfied) to 5 or 7 (most satisfied). A total score is then summed for each domain on the following scales: effectiveness 1-21, side effects 1-20, convenience 1-21, and global satisfaction 1-17. Lower total scores in each domain indicate dissatisfaction with the study medication and higher total scores indicate satisfaction.
Time Frame: At Baseline and Week 16
Population: as for outcome 20
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 28
score on a scale
  Effectiveness: number analyzed (Participants) | 24
  Effectiveness | 4.76 [-28.6 to 42.9]
  Side Effects: number analyzed (Participants) | 10
  Side Effects | 5.00 [-50.0 to 35.0]
  Convenience: number analyzed (Participants) | 25
  Convenience | -4.76 [-52.4 to 28.6]
  Global Satisfaction: number analyzed (Participants) | 25
  Global Satisfaction | 0.00 [-47.1 to 35.3]

23. Secondary Outcome: Improvement From Baseline in Clinical Risk Category
Description: 6MWD low risk: >440 m, intermediate risk: 165-440 m, high risk: <165 m; NT-proBNP low risk: <300 ng/L, intermediate risk: 300-1400 ng/L, high risk: >1400 ng/L; WHO FC: low risk: I or II, intermediate risk: III, high risk: IV; and Right Atrial Area: low risk: <18 cm², intermediate risk: 18-26 cm², high risk: >26 cm². Moving from a higher risk category to a low risk category was considered "improved;" moving from a lower risk category to a higher risk category was considered "worsened."
Time Frame: At Baseline and Week 16
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 29
Participants
  6MWD: number analyzed (Participants) | 27
  6MWD: Improved | 4
  6MWD: Worsened | 1
  6MWD: No Change | 22
  NT-proBNP: number analyzed (Participants) | 28
  NT-proBNP: Improved | 11
  NT-proBNP: Worsened | 1
  NT-proBNP: No Change | 16
  WHO FC: number analyzed (Participants) | 28
  WHO FC: Improved | 11
  WHO FC: Worsened | 1
  WHO FC: No Change | 16
  Right Atrial Area: number analyzed (Participants) | 23
  Right Atrial Area: Improved | 8
  Right Atrial Area: Worsened | 1
  Right Atrial Area: No Change | 14

24. Secondary Outcome: Achievement of Low Risk Category in Clinical Parameters
Description: Low risk categories for the 4 selected parameters were: 6MWD >440 m, serum NT-proBNP <300 ng/L, WHO FC I or II, and right atrial area <18cm². The rows of the table indicate the count of participants that were in the low risk category for the parameter at Week 16.
Time Frame: At Week 16
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 29
Participants
  6MWD: number analyzed (Participants) | 27
  6MWD | 10
  NT-proBNP: number analyzed (Participants) | 28
  NT-proBNP | 19
  WHO FC: number analyzed (Participants) | 28
  WHO FC | 24
  Right Atrial Area: number analyzed (Participants) | 23
  Right Atrial Area | 14

25. Secondary Outcome: Overall Achievement
Description: The percentage of subjects that ended the study in achievement Class 1 (either achieved an Orenitram dose of ≥4 mg TID [or TDD of 12 mg] at Week 16 or a dose of ≥0.057 mg/kg TID [or a TDD of 0.171 mg/kg] for subjects <70 kg), Class 2 (achieved a prescribed Orenitram dose ≥2 mg TID and <4 mg TID [or a TDD ≥6 mg and <12 mg] at specific visit, with at least 2 of the following 3 clinical parameters: 6MWD increase by ≥10% or ≥30 m from baseline, serum NT-proBNP reduction >30% from baseline, or WHO FC I or II), or Class 3 (were not Class 1 or Class 2, or with class undetermined).
Time Frame: At Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 29
Participants
  Class 1 | 23
  Class 2 | 2
  Class 3 | 4

26. Secondary Outcome: Transition and Maintenance of Orenitram Therapy
Description: The percentage of subjects that transitioned to oral treprostinil at any dose and were maintained on therapy at Week 16 (considered a "successful" result).
Time Frame: At Week 16
Population: Per-protocol Population. Only Subjects with Baseline and Week 16 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
Number analyzed (Participants) | 29
Participants | 28

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were captured from when the subject signed the informed consent form until the subject completed the study or was withdrawn from the study, up to 20 weeks.
Description: AEs were followed until either resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, or for at least 4 weeks if the AE extended beyond the final study visit (Week 16). All serious adverse events (SAEs) that occurred during the study were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 4 weeks after completion of the final study visit.
Arm/Group | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil (N=35)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic embolus (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous/Subcutaneous Treprostinil; Oral Treprostinil (N=35)
Nausea (Gastrointestinal disorders) | 25 (27)
Diarrhoea (Gastrointestinal disorders) | 21 (22)
Vomiting (Gastrointestinal disorders) | 15 (17)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 30 (33)
Dizziness (Nervous system disorders) | 7 (10)
Syncope (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 14 (14)
Infusion site pain (General disorders) | 9 (9)
Pain (General disorders) | 9 (9)
Oedema peripheral (General disorders) | 6 (6)
Infusion site irritation (General disorders) | 5 (5)
Chills (General disorders) | 2 (2)
Infusion site swelling (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 18 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (17)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 20 (20)
Hot flush (Vascular disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Infusion site infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Device dislocation (Product Issues) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT03497689/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03497689/SAP_001.pdf